CLINICAL TRIAL: NCT03385460
Title: Delivery of Intravesical Botulinum Toxin A Using Low Energy Shock Waves in Treatment of Overactive Bladder: A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed Nageib, Msc, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOTOX-SWL
Record Dates: First submitted 2017-12-13; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Overactive Bladder; Botulinum Toxin; Intravesical; ESWL
Keywords: Overactive bladder; Botulinum Toxin; low energy shock waves; Intravesical
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESWL BOTOX (Experimental): Each patient will be subjected to Low Energy Shock Waves.The target dose of low energy shock waves will be 3000 shock delivered into SP region in 3 horizontal points at SP transverse crease . all patients will be catheterized using nylaton catheter 16 ch, the study group will be injected with 100 IU botulinium toxin A. vial will be dissolved in saline half of the estimated bladder capacity. All patients will be kept for 2 hours without micturation giving a chance of BOTOX absorption .
  Interventions: Other: ESWL BOTOX

INTERVENTIONS:
Other: ESWL BOTOX — ESWL after intrravesical BOTOX

SUMMARY:
We hypothesize that LESWs might temporarily increase urothelial permeability and facilitate delivery of intravesical botulinum toxin without the need for injection.

DETAILED DESCRIPTION:
High energy extracorporeal shock wave thrapy has been used to disintegrate urolithiasis for 30 years (Chaussy et al., 1982). Low energy shock wave LESWs are used clinically to improve tissue regeneration at tendon- bone junctions (Wang et al., 2003) , ischemic cardiovascular disorders (Dimeglio et al., 2012) and erectile dysfunctions (Vardi et al., 2012).

Furthermore, shock waves have been shown to temporarily increase tissue permeability (Lauer et al., 1997, Kodama et al., 2002) and increase mediated molecular and drug delivery into cells without consequent cytotoxicity. Kodama et al., 2002 suggested that shock waves could cause shear force generated by the movement of liquid relative to cells to temporarily affect the permeability of the plasma memberance. Shock waves can deliver molecules to 2,000,000 molecular weight into the cystoplasm of cells without toxicity (Lauer et al., 1997).

Instillation of drugs in the bladder provides the opportunity to locally increase drug concentration with a low risk of systemic side effects (Kuo et al., 2010, Hsu et al., 2013). Intravesical pharmacotherapy has been used to treat refractory overactive bladder and interstitial cystitis/ painful bladder syndrome (smith et al., 2004; Grannantoni et al., 2008; Boy et al., 2006). However, drug delivery to bladder tissues by intravesical route is constrained by urothelial impermeability. The watertight barrier is generally located at the umbrella cells, which are the superficial layers of bladder epithelium augmented by glycosaminoglycans and uroplakins (Hsu et al., 2013; Birder et al., 2005).

Transient permeabilization of cell membranes accomplished by shock waves can deliver macromolecular drugs in the bladder without toxicity (Lower et al., 1997; Kodama et al., 2002).

Chuang et al., (2016) demonstrated that contrast enhanced MRI can detect increased rat bladder permeability after LESWs. Recently, Towner et al (2015) reported increased urothelial permeability and contrast leakage on bladder MRI after intravesical promtamine sulfate instillation.

Chen et al., (2014) found that LESWs treatment 3 and 24 hours after cyclophosphamide administration could attenuate cyclophosphamide induced acute cystitis in rats by decreasing inflammation and oxidative stress.

In a recent study, Chuang et al., (2016) investigated the feasibiblity of using LESWs for intravesical botulinum toxin A delivery. They evaluated the efficacy for acetic acid included bladder hyperactivity in rats. They concluded that LESWs increased urothelial permeability, facilitate intravesical botulinum toxin A delivery and block acetic acid included hyperactive bladder. These results support LESWs as a promising method to deliver botulinum toxin A without the need for injection.

Overactive bladder (OAB) is a condition characterized by presence of urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence [UUI], in the absence of urinary tract infection (UTI) or other obvious pathology (Haylen BT et al 2010). OAB is a common problem that impair the quality of life (QOL).The prevalence of OAB ranged from 11.8% in a population-based survey conducted across five European countries ( Irwin DE et al, 2008 ) to 16.9% according to Epidemiological studies from North America and the prevalence increases with age rising to 30.9% in those over the age of 65 years.( Stewart WF et al 2001) Treatment goals are to reduce the occurrence of bothersome symptoms, and provide beneﬁts that are perceived by patients as meaningful (Brubaker L et al, 2006). Several treatment options are available for OAB including bladder and behavioral training , pharmacologic treatment , and surgical therapies (Wein AJ et al, 2006).

Antimuscarinics are well established as pharmacotherapy for reducing OAB symptoms and improving QOL (Andersson KE et al, 2009). However, their use is limited in some patients by insufficient response to treatment "refractory OAB", or intolerable side effects such as dry mouth ,blurred vision, constipation, and cognitive impairment (Benner JS et al, 2010).

After a trial of pharmacotherapy, if the patient has not had an adequate improvement in symptoms, intra-vesical injection of Botox (BTX) can be offered as the next step. Botulinum toxin (BTX) is a neurotoxin, it contains a heavy chain that binds to the presynaptic terminal of the neuromuscular junction , and this then acts by inhibiting the release of acetylcholine from the presynaptic vesicles at the axon terminal of the motor end plate , that then result in the muscle that is innervated becoming ﬂaccidly paralyzed. BTX is available in different preparations, each of which is a distinct chemical entity. The current commercially utilized type is BTX type A.

Currently, there is cumulative data supporting use of BTX in cases of refractory Deturosr overactivity. Intradetrusal injection of BTX is followed by a significant improvements in the number of voiding episodes over 24 h, incontinence episodes, urodynamic variables and quality-of -life scores (Mangera A et al, 2011). There is a reduction in episodes of urgency and incontinence by 80% and 60%, respectively. The efficacy peaks at 4 weeks ,with the effect lasting typically up to 9 months , and repeated treatment efficacy has been shown in up to 10 treatment cycles. Patients should be counseled about the risk of an increased postvoid residual volume, occurring in 20-40% of individuals, and the need to use self-catheterization, with the attendant risk of UTI (14-40%) (Mangera A et al, 2011). The risk of general muscular weakness is considered very rare.

ELIGIBILITY:
Inclusion Criteria:

* OAB refractory to treatment with antimuscarinics for 2 months

Exclusion Criteria:

* Sensitivity to botox
* Neurogenic detrusor overactivity
* Active UTI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 10 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Intravesical Botulinum Toxin A Delivery Using Low Energy Shock Waves for management of OAB: Pressure flow urodynamics measured in cm/H2O | 1 year
  pressure flow urodynamics will be measured in cm/H2O

SECONDARY OUTCOMES:
Impact of the new technique on the quality of life based on QOL score | 1 year
  OAB symptoms score

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and nephrology center, Al Mansurah, Egypt